CLINICAL TRIAL: NCT06295627
Title: The Analysis of Factors Causing Indwelling Urinary Catheter-related Infections in ICU Patients and Their Nursing Strategies
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2024-115-01
Record Dates: First submitted 2024-02-05; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Catheter-associated Urinary Tract Infection
Keywords: ICU; Catheter-associated; Factors; NursingCountermeasures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infected group: The infection group consisted of patients with urinary tract infection (13 cases)
  Interventions: Other: There were no interventions in retrospective analysis
- Non-infected group: Non-infection group The first group consisted of patients without urinary tract infection (278 cases)
  Interventions: Other: There were no interventions in retrospective analysis

INTERVENTIONS:
Other: There were no interventions in retrospective analysis — A retrospective analysis method was used to analyze the causes of catheter-related urinary tract infection and the infecting bacteria of the two groups of patients. A single factor analysis was performed on various factors and other related factors, and corresponding nursing strategies were summarized and proposed.

SUMMARY:
To explore the analysis of factors causing indwelling urinary catheter-related infections in ICU patients and their nursing strategies, and to provide reference for clinical nursing work. 291 patients with indwelling urinary catheters in the second area of ICU of our hospital from January 1, 2023 to September 30, 2023 were selected as research subjects. They were divided into infection group and non-infection group according to the presence or absence of urinary tract infection. Non-infection group The first group consisted of patients without urinary tract infection (278 cases), and the infection group consisted of patients with urinary tract infection (13 cases). A retrospective analysis method was used to analyze the causes of catheter-related urinary tract infection and the infecting bacteria of the two groups of patients. A single factor analysis was performed on various factors and other related factors, and corresponding nursing strategies were summarized and proposed.

ELIGIBILITY:
Inclusion Criteria:

* Age > 14 years
* Patients with indwelling urinary tube during hospitalization
* Length of stay in ICU > 48h
* Complete hospitalization data

Exclusion Criteria:

* Had urinary tract infection before hospitalization
* Indwelling catheter < 72h
* Severe liver and kidney failure and death within 48 hours of admission

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 291 patients with indwelling urinary catheters in the second area of ICU of our hospital from January 1, 2023 to September 30, 2023 were selected as research subjects.
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
How many patients in the infected group and how many patients in the non-infected group had bladder irrigation | 2023.1.1-2023.9.30
  Bladder irrigation is easy to damage the drainage tightness of urinary system and increase the risk of infection. Frequent irrigation is easy to lead to urinary tract infection.SPSS27.0 software was used to analyze and process the bladder irrigation data of the two groups of patients.
How many patients in the infected group and how many patients in the non-infected group were given enema | 2023.1.1-2023.9.30
  Patients with increased frequency of stool after enema, fecal incontinence or diarrhea are at risk of retrograde infection caused by fecal contamination of the urethral opening.SPSS27.0 software was used to analyze and process the enema data of the two groups of patients.
How many times the indwelling catheter was changed in patients in the infected group and patients in the non-infected group respectively | 2023.1.1-2023.9.30
  Indwelling catheter can easily lead to urethral mucosa injury, and the urethral mucosa is damaged repeatedly by repeated intubation, and the normal physiological barrier is damaged and the risk of urinary tract infection is increased.SPSS27.0 software was used to analyze and process the data of the number of indwelling catheters in the two groups
How many patients in the infected group and the non-infected group had co-diabetes | 2023.1.1-2023.9.30
  Urinary tract infection is the most common infection in patients with diabetes, and the high blood sugar state of the body helps bacteria colonize and proliferate.The combined diabetes data of the two groups were analyzed and processed using SPSS27.0 software.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong, China